CLINICAL TRIAL: NCT03436511
Title: Burden of Disease Among Patients With Eosinophilic COPD in Spain: Multicentre Observational Study
Brief Title: Burden of Disease Among Subjects With Eosinophilic Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Oblikue Consulting (Unknown)
Responsible Party: Sponsor
Other Study IDs: 206555
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Health resource utilization; Eosinophilic COPD; Mepolizumab
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with COPD: Subjects with a COPD diagnosis confirmed with a post-bronchodilator Forced Expiratory Volume in 1 second/Forced Vital capacity <70% recorded at any time in the medical record who have a qualifying peripheral blood eosinophil test recorded in the 3 months prior to the inclusion visit attend to a routine follow-up visit during the inclusion period, fulfill the inclusion/exclusion criteria and provide informed consent to participate, will be included in this study.

SUMMARY:
This observational study is designed to more specifically describe the burden of the disease and the use of healthcare resources of subjects with eosinophilic COPD that may be eligible in the future for a biologic treatment. Subjects who attend a routine follow-up visit and fulfill the inclusion/exclusion criteria defined provide a signed informed consent will be invited by the investigator to participate in this study. Subjects will be recruited in hospital Pulmonology Services across Spain. It is planned to include approximately 20 centers. To select the final participating centers, a feasibility study has been carried out in approximately 50 potential participating centers. It has been estimated that each investigator will include 18 subjects during the 4-month inclusion period. Total 354 subjects will be required: 250 subjects with an eosinophil level >=150 cells per microliter and 104 subjects with an eosinophil level <150 cells per microliter. The study inclusion period will be 4 months (expected to be from November 2017 to March 2018) and the retrospective data collection period will be 12 months prior to the inclusion visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes aged >=40 years.
* Subjects with a COPD diagnosis confirmed with a post-bronchodilator Forced Expiratory Volume in 1 second/Forced Vital capacity <70% recorded at any time in the medical record.
* Subjects with a history of smoking (current or past) >=10 pack-years.
* Subjects who have a qualifying peripheral blood eosinophil test recorded in the 3 months prior to the inclusion visit. If the subject has several eosinophil test recorded in this period, the one closest to the inclusion visit determined in the stable phase should be selected; if it is not available, the record closest to the inclusion visit will be selected, even if it has been determined during an exacerbation. If no records are available, the subject will be invited to perform the test at the inclusion visit.
* Subjects currently exposed to inhaled triple maintenance therapy, defined as at least one overlapping prescription of an ICS with a LABA and with a LAMA in 2 or 3 inhaler devices, without more than 30 days of separation between prescriptions.
* Subjects who have experienced >=2 moderate exacerbations or >=1 severe exacerbation in the 12 months prior to the inclusion visit. Moderate exacerbation is defined as an exacerbation requiring antibiotics and/or oral corticosteroids or requiring an emergency visit <24 hours (without hospitalization). Severe exacerbation is defined as an exacerbation requiring hospitalization.
* Subjects who consent to participate in the study by signing the subjects written informed consent form.

Exclusion Criteria:

* Subjects without a qualifying peripheral blood eosinophil test recorded in the 3 months prior to the inclusion visit and who refuse to perform the test during the inclusion visit.
* Subjects treated with oral corticosteroids continuously during the 12 months prior to the inclusion visit.
* Subjects with a diagnosis of Churg-Strauss disease, hypereosinophilic syndrome, allergic bronchopulmonary aspergillosis or other conditions that result in increased eosinophil levels independently of COPD.
* Subjects with oncologic disease undergoing treatment or with advanced oncologic disease (without possibility of remission), terminal subjects and/or subjects receiving palliative care.
* Cognitively impaired subjects who are not able to understand or complete the informed consent and HRQoL questionnaires.
* Subjects who have participated in an interventional clinical trial during the 12 months prior to the inclusion visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who attend a routine follow-up visit and who fulfill inclusion/exclusion criteria will be invited by the investigator to participate in the study. The study inclusion period will be four months (from November 2017 to March 2018) and the retrospective data collection period will be 12 months prior to the inclusion visit.
Sampling Method: Non-Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects requiring COPD maintenance treatment and rescue medication | 12 months prior to the inclusion visit
  Subjects currently exposed to inhaled triple maintenance therapy, defined as at least one overlapping prescription of an inhaled corticosteroid (ICS) with a long-acting beta2-agonist (LABA) and with a long-acting muscarinic antagonist (LAMA) in 2 or 3 inhaler devices, without more than 30 days of separation between prescriptions along with rescue medication use will be analyzed.
Number of subjects with moderate and severe exacerbations | 12 months prior to the inclusion visit
  Subjects who have experienced >=2 moderate exacerbations or >=1 severe exacerbation in the 12 months prior to the inclusion visit. Moderate exacerbation is defined as an exacerbation requiring antibiotics and/or oral corticosteroids or requiring an emergency visit <24 hours (without hospitalization). Severe exacerbation is defined as an exacerbation requiring hospitalization.
Number of subjects with COPD-related scheduled and unscheduled primary and secondary care visits | 12 months prior to the inclusion visit
  Subjects with COPD-related scheduled and unscheduled primary and secondary care visits will be analyzed.
Number of subjects with COPD-related emergency visits to primary care and hospital | 12 months prior to the inclusion visit
  Subjects with COPD-related emergency visits to primary care and hospital will be analyzed.
Number of subjects with COPD-related hospitalizations | 12 months prior to the inclusion visit
  Subjects with COPD-related hospitalizations will be analyzed.
Number of days of hospitalizations | 12 months prior to the inclusion visit
  The number of days of hospitalization for subjects will be analyzed.
Number of subjects with COPD-related complementary tests | 12 months prior to the inclusion visit
  Subjects with COPD-related complementary tests will be analyzed.
Number of subjects with COPD-related days-off work | 12 months prior to the inclusion visit
  Subjects with COPD-related days-off work will be analyzed.

SECONDARY OUTCOMES:
Subjects age as a measure of sociodemographic characteristics | 4 months (inclusion period)
  Age will be recorded for descriptive analysis of the sociodemographic characteristics of the subjects participating in the study. A threshold of >=150 cells/microliter will be considered to determine a high level of eosinophil's, so only subjects meeting this criterion will be included in the analysis.
Number of subjects with different gender | 4 months (inclusion period)
  Gender will be recorded for descriptive analysis of the sociodemographic characteristics of the subjects participating in the study. A threshold of >=150 cells/microliter will be considered to determine a high level of eosinophil's, so only subjects meeting this criterion will be included in the analysis.
Number of subjects with different sociodemographic variables | 4 months (inclusion period)
  Subjects with different educational level, employment status, monthly net income will be recorded for descriptive analysis of the sociodemographic characteristics of the subjects participating in the study A threshold of >=150 cells/microliter will be considered to determine a high level of eosinophil's, so only subjects meeting this criterion will be included in the analysis.
Number of subjects with abnormal clinical variables | 4 months (inclusion period)
  Clinical variables comprising weight, height, body mass index (self-calculated), smoking history, Charlson comorbidity index, diagnosis of asthma will be assessed for abnormalities. A threshold of >=150 cells/microliter will be considered to determine a high level of eosinophil's, so only subjects meeting this criterion will be included in the analysis.
Number of subjects with abnormal COPD related variables | 12 months prior to the inclusion visit
  COPD variables comprising COPD diagnosis date, pulmonary function with bronchodilator test, modified Medical Research Council (mMRC) dyspnea scale, clinical phenotypes according to Spanish COPD Clinical Guidelines (GesEPOC) criteria will be assessed for abnormalities. A threshold of >=150 cells/microliter will be considered to determine a high level of eosinophil's, so only subjects meeting this criterion will be included in the analysis.
Number of subjects with abnormal blood cell count | 12 months prior to the inclusion visit
  Peripheral blood eosinophil count, peripheral blood neutrophil count, peripheral blood leukocyte count, fibrinogen and red cell distribution width will be assessed for abnormalities.
COPD Assessment Test (CAT) score as a measure of Health Related Quality of Life (HRQoL) | 4 months (inclusion period)
  The CAT questionnaire is a COPD-specific questionnaire that measures the impact of the disease on HRQoL and allows symptoms to be described. It consists of 8 items, which yield a score range from 0 to 40, 0 representing the lowest impact on HRQoL and 40 the maximum impact.
EuroQOL five dimensions five level (EQ-5D-5L) score as a measure of HRQoL | 4 months (inclusion period)
  The EQ-5D-5L is a preference-based generic HRQoL questionnaire, consisting on five health dimensions (mobility, personal care, daily activities, pain/discomfort and anxiety/depression), divided in five levels of severity (no problems, slight problems, moderate problems, severe problems and extreme problems). It included also a visual analogue scale (VAS) in which respondents are asked to evaluate their overall health status on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (3):
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Valencia